CLINICAL TRIAL: NCT04313868
Title: A Phase 1 Dose Escalation Trial to Evaluate the Safety, Pharmacokinetics, and Pharmacodynamics of GEN2 in Refractory Patients With Primary Hepatocellular Carcinoma or Tumors Metastatic to the Liver
Brief Title: GEN2 Directed Cancer Immunotherapy Trial
Acronym: GEN2
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GenVivo, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: EPB-002
Record Dates: First submitted 2020-01-15; First posted 2020-03-18 (Actual); Last update posted 2024-11-06 (Actual); Status verified 2024-11

CONDITIONS: Hepatocellular Carcinoma; Metastatic Cancer
Keywords: Liver Metastasis; Liver Cancer
MeSH Terms: conditions — Carcinoma, Hepatocellular; Neoplasm Metastasis; Liver Neoplasms

STUDY DESIGN:
Intervention Model Description: Dose Escalation Trial
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Phase 1A.1: Peripheral IV (Experimental): GEN2 is administered in repeating three week cycles. On week one, GEN2 is given intravenously on three consecutive days and the presence of the HSV-TK-m2 expression is monitored by [18F]FHBG PET scanning after 3 to 8 days. Valganciclovir dosing is initiated on day 7 to 9 for 5 days. An approximately one week drug holiday follows.
  Interventions: Drug: GEN2 (HSV-Thymidine Kinase-m2 and hGM-CSF Genes)
- Phase IA.2: Hepatic Artery Infusion (Experimental): GEN2 is administered in repeating three week cycles. On week one, GEN2 is given as a single hepatic artery infusion (HAI) on two successive days and the presence of the HSV-TK-m2 expression is monitored by [18F]FHBG PET scanning after 3 to 8 days. Valganciclovir dosing is initiated on day 7 to 9 for 5 days. An approximately one week drug holiday follows.
  Interventions: Drug: GEN2 (HSV-Thymidine Kinase-m2 and hGM-CSF Genes)
- Phase IA.3: Intratumoral Injection (Experimental): GEN2 is administered in repeating three week cycles. On week one, GEN2 is given via injection directly into the tumor lesions on one day and the presence of the HSV-TK-m2 expression is monitored by [18F]FHBG PET scanning after 3 to 8 days. Valganciclovir dosing is initiated on day 7 to 9 for 5 days. An approximately one week drug holiday follows.
  Interventions: Drug: GEN2 (HSV-Thymidine Kinase-m2 and hGM-CSF Genes)

INTERVENTIONS:
Drug: GEN2 (HSV-Thymidine Kinase-m2 and hGM-CSF Genes) — GEN2 is an investigational drug combining cytotoxic and immunotherapy.

SUMMARY:
Phase 1, non-randomized, open label dose escalation clinical trial evaluating the safety of GEN2 in participants with primary & metastatic liver tumors.

DETAILED DESCRIPTION:
This clinical trial will be divided into two phases: Phase IA in which the dose, route, and schedule of the GEN2 administration is determined and Phase IB which is designed to explore the activity of GEN2 in patients of a defined or several defined tumor types and stages based on the Phase IA data of GEN2.

Phase IA is divided into three routes of administration: (a) Phase 1A.1 which explores peripheral IV infusion; (b) Phase IA.2 which investigates hepatic arterial infusion and (c) Phase IA.3 which examines intratumoral delivery.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of histologically documented, advanced stage, primary or metastatic adult solid tumor(2) in the liver that are refractory to standard therapy or for which no curative standard therapy exists.
* Evidence of radiographically measurable or evaluation disease on a baseline PET-CT scan.
* All acute toxic effects of any prior radiotherapy, chemotherapy, or surgical procedures must have resolved to National Cancer Institute (NCI) Common Toxicity Criteria (CTC) (Version 4.03) Grade < 1.
* Patient must be legally considered an adult in the country in which they are participating in the study.
* Last dose of antineoplastic therapy, except for hormonal therapy, must be > 21 days. External beam radiotherapy must have been <25% bone marrow-containing skeleton.
* Patients may be Hepatitis B and C positive.
* Patients may have intracranial metastases of any number if they have been brain irradiated and stable for 6 weeks. Patients may be taking anti-seizure medicines but must not be on steroids. Last dose of steroids must be >7 days.
* Karnofsky performance status must be > or = 70
* Childs-Pugh Classification Score of 7 or less
* Life Expectancy of at least 3 months
* Patients must be able to travel to alternate medical center for PET/CT scans, if necessary.
* Meet the required baseline laboratory data
* Signed informed consent indicating that they are aware of the neoplastic nature of their disease and have been informed of the procedures to be followed, the experimental nature of the therapy, alternatives, potential benefits, side effects, risks and discomforts.
* Willing and able to comply with scheduled visits, treatment plan, and laboratory tests.

Exclusion Criteria:

* Concurrent therapy with anticancer agent including any other investigational agent.
* Existing intracranial edema or CVA within 6 months of screening
* Pregnant or breast-feeding women. Female patients must agree to use effective contraception, must be surgically sterile or must be post-menopausal. Male patients must agree to use effective contraception or be surgically sterile. The definition of effective contraception will be based on the judgment of the Investigator or a designated associate. All at-risk female patients must have a negative pregnancy test within 7 days prior to start of the study treatment.
* Clinically significant cardiac disease (New York Heart Associate, Class III or IV)
* Dementia or altered mental status that would prohibit informed consent.
* Other severe, acute, or chronic medical or psychiatric condition or laboratory abnormality that may increase the risk associated with study participation of study results and, in the judgment of the Investigator, would make the patient inappropriate for this study.
* Known side effects to antivirals in the ganciclovir class
* Patients who are known to be HIV positive.
* Patients must not be taking steroids at the time of screening. Last dose of steroids must be >7 days.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2014-06-13 (Actual); Primary Completion 2023-12-12 (Actual); Study Completion 2023-12-12 (Actual)

PRIMARY OUTCOMES:
Maximum Tolerated Dose (MTD) | First 3 weeks of GEN2 Administration
  The MTD is the defined as the highest dose level at which, at most, one patient experiences a DLT.
Dose Limiting Toxicity (DLT) | First 3 weeks of GEN2 Administration
  * Grade 4 neutropenia
  * Grade 4 thrombocytopenia;
  * Grade 3 or greater nausea and/or vomiting despite the use of adequate/maximal medical intervention and/or prophylaxis;
  * Any Grade 3 or greater non-hematological toxicity (except Grade 3 injection site reaction, alopecia, fatigue);
  * Retreatment delay of more than 3 weeks due to delayed recovery from a toxicity related to treatment with GEN2;
  * Grade 3 or greater allergic (hypersensitivity) reaction despite the appropriate use of premedications (defined within the CTC as "Prolonged" (e.g., not rapidly reponsive to symptomatic medication and/or brief interruption of infusion); recurrence of symptoms following initial improvement; hospitalization indicated for clinical sequelae (e.g., renal impairment, pulmonary infiltrates).
Recommended Phase 2 Dose (RP2D) | First 3 weeks of GEN2 Administration
  The RP2D will be administered for Phase 1B. It is determined when the accelerated phase ends for Phase IA and the dose assignment for a new patient in the standard dose escalation will follow a modified Fibonacci scheme. If a modified Fibonacci has already been used, the RP2D will be explored from the remaining intervals between the dose which had no DLTs and the Maximum Administered Dose (MAD).
Number of participants with treatment-related adverse events as assessed by CTCAE v4.0 | Treatment Initiation until 30 days after last dose of GEN2
  Each Adverse Event is to be classified by the Investigator as serious or non-serious. The classification of the gravity of the event determines the reporting procedures to be followed.

SECONDARY OUTCOMES:
Plasma pharmacokinetics of GEN2 | During Week 1 of Cycle 1, Cycle 2 & Cycle 6 (each cycle is 28 days)
  GEN2 PK Cmax is dose proportional.
HSV-TK-m2 protein expression from GEN2 via serial [18F]FHBG PET and/or SPECT imaging | Day 3-8 of GEN2 Treatment
  Identify number of participants with positive [18F] FHBG scan
Preliminary Evidence of anti-tumor activity of GEN2 | Week 9 and every 6 weeks thereafter through study completion, an average of 8 months.
  Measure of anti-tumor efficacy based on objective tumor assessments made according to the irRECIST 1.1
Clinical research testing for antibodies to retrovector gp70 env, replication-competent retrovirus in peripheral blood lymphocytes (PBLs); vector integration into genomic DNA of PBLs, and circulating hGM-CSF protein | Cycle 1, Cycle 2, Cycle 6, after 6th month on treatment, annually thereafter
  No replication-competent retrovirus. No vector integration into genomic DNA of PBLS. No GM-CSF detectable in patients after GEN2 administration

CONTACTS AND LOCATIONS:
Overall Officials: Priscilla B Caguioa, MD, Principal Investigator — St. Luke's Medical Center - Quezon City; Maria Belen E Tamayo, MD, Principal Investigator — Makati Medical Center; John P Querol, MD, Principal Investigator — The Medical City; Necy S Juat, MD, Principal Investigator — National Kidney and Transplant Institute
Locations (4):
- Philippines (4):
  - Makati Medical Center, Makati City
  - The Medical City, Pasig
  - National Kidney and Transplant Institute, Quezon City
  - St. Luke's Medical Center, Quezon City